CLINICAL TRIAL: NCT00438737
Title: Randomized Phase II Trial Evaluating the Feasibility and Tolerance of the Combination of FOLFOX With Cetuximab and the Combination of FOLFOX With Cetuximab and Bevacizumab as Perioperative Treatment in Patients With Resectable Liver Metastases From Colorectal Cancer
Brief Title: Cetuximab, Leucovorin, Oxaliplatin, and Fluorouracil With or Without Bevacizumab in Treating Patients With Resectable Liver Metastases From Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000530116; EORTC-40051; EUDRACT-2005-002825-29; EU-20776
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2007-09

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Cetuximab; Fluorouracil; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Biological: bevacizumab
Biological: cetuximab
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor.Drugs used in chemotherapy, such as leucovorin, oxaliplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with combination chemotherapy and bevacizumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This randomized phase II trial is studying the side effects and how well giving cetuximab together with leucovorin, oxaliplatin, and fluorouracil works with or without bevacizumab in treating patients with resectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety and activity of neoadjuvant and adjuvant cetuximab, leucovorin calcium, oxaliplatin, and fluorouracil with vs without bevacizumab in patients with resectable liver metastases secondary to colorectal cancer.

OUTLINE: This is an open-label, randomized, multicenter study. Patient are stratified according to participating center and planned liver resection (major [≥ 3 segments] vs minor [< 3 segments]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive leucovorin calcium IV over 2 hours and oxaliplatin IV over 2 hours on day 1 and fluorouracil IV over 46 hours (FOLFOX) beginning on day 1. Patients also receive cetuximab IV over 1-2 hours on days 1 and 8. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Between 3-5 weeks after completion of FOLFOX and cetuximab, patients undergo liver resection. Beginning between 4-8 weeks after surgery, patients receive another 6 courses of FOLFOX and cetuximab as in neoadjuvant therapy.

* Arm II: Patients receive FOLFOX and cetuximab as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 14 days for 6 courses* in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients do not receive bevacizumab during course 6

Between 3-5 weeks after completion of FOLFOX, cetuximab, and bevacizumab, patients undergo liver resection. Beginning between 4-8 weeks after surgery, patients receive another 6 courses of FOLFOX, cetuximab, and bevacizumab as in neoadjuvant therapy.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for at least 3 years.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic colorectal cancer, meeting all of the following criteria:

  * Metachronous or synchronous liver metastases

    * Metastases potentially completely resectable

      * No requirement for resection combined with cryotherapy or radiofrequency ablation
  * Must have undergone complete resection (R0) of the primary tumor within the past 4 weeks
* Measurable liver metastases
* No evidence of extrahepatic disease

  * 1 or 2 resectable lung metastases allowed

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 9 g/dL
* WBC > 3,000/mm³
* Creatinine < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* AST and ALT < 5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant proteinuria (i.e., protein > 500 mg/24-hour urine collection)
* No known allergy to any of the study drugs (including excipients) or any related compound, including hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* No bleeding diathesis or coagulopathy
* No peripheral neuropathy > grade 1
* No serious nonhealing wound, ulcer, or bone fracture
* No clinically significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension
  * New York Heart Association class II-IV congestive heart failure
  * Unstable angina pectoris within the past 12 months
  * Peripheral vascular disease ≥ grade 2
  * Serious cardiac arrhythmia requiring medication
  * Myocardial infarction within the past 12 months
  * Cerebrovascular accident or transient ischemic attack within the past 12 months
* No symptomatic diverticulitis or known gastroduodenal ulceration
* No significant traumatic injury within the past 4 weeks
* No known alcohol or drug abuse
* No psychological, familial, social, or geographical condition that would preclude study compliance
* No other significant disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for metastatic disease
* At least 1 month since prior major surgical procedure or open biopsy
* More than 30 days since prior participation in another clinical study
* Prior adjuvant chemotherapy for primary cancer allowed provided the following criteria are met:

  * At least 12 months since prior oxaliplatin-containing adjuvant therapy
  * No persistent neuropathy
* No prior therapy targeting the epidermal growth factor receptor or vascular endothelial growth factor (VEGF)/VEGF receptor
* No concurrent regular use of acetylsalicylic acid (> 325 mg/day) or other nonsteroidal anti-inflammatory drugs
* No concurrent full-dose anticoagulation
* No concurrent prophylactic hematopoietic growth factors
* No concurrent allopurinol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Response rate (preoperative response rate)
Safety (rate of perioperative safety findings)

SECONDARY OUTCOMES:
Progression-free survival
Pathological resection rate
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Nordlinger, MD — Hopital Ambroise Pare
Locations (1):
- Hopital Ambroise Pare, Boulogne, France